CLINICAL TRIAL: NCT03135080
Title: The Effect of Long-Term HEAD START Training on Surgical Skill Levels
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: International Agency for the Prevention of Blindness (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 17-0423
Record Dates: First submitted 2017-04-11; First posted 2017-05-01 (Actual); Last update posted 2018-03-15 (Actual); Status verified 2018-03

CONDITIONS: Trichiasis; Surgery
MeSH Terms: conditions — Trichiasis | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: All study participants will have their skill levels on live surgery evaluated at the end of surgical training and again at the start of the surgical season, approximately 6 months later. Fifteen trainees will participate in long-term HEAD START practice and receive feedback throughout this break during the rainy season when surgical activity is low. An additional 15 individuals will be selected for the trainer to assess their skill levels on live surgery at the end of training and again at the start of the surgical season this fall but will not receive additional surgical practice.
Who Masked: Outcomes Assessor
Masking Description: At the end of the rainy season, an independent examiner (not involved in the HEAD START evaluations) will assess the first 1-2 surgeries of the season of all study participants. The assessor will not know whether surgeons had participated in the long-term HEAD START training over the rainy season.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Long-term HEAD START Training (Experimental): Fifteen surgeons will participate in long-term HEAD START practice once live surgical training is complete. Each week the participant will complete 2 surgeries on the HEAD START device and mark the surgery number on the cartridge. Monthly, the participant will send the accumulated cartridges to Addis for review by a senior trichiasis surgery trainer. The trainer will evaluate the cartridges and then will discuss his/her impression of the surgeries with the participant during a regular monthly call. He/she will also note the findings on a standardized form. Practice will continue for approximately 4-6 months, depending on the length of the rainy season and time of enrollment.
  Interventions: Other: Long-Term HEAD START Training
- Standard of Care (Active Comparator): Once live surgical training is complete, fifteen surgeons will commence live surgery without supervision until the rainy season begins. Then they will break for the rainy season, per the typical practice. The trainer will assess their skill levels on live surgery at the end of training and again at the start of the surgical season in the fall.
  Interventions: Other: Standard of Care

INTERVENTIONS:
Other: Long-Term HEAD START Training — The Human Eyelid Analogue Device for Surgical Training And skill Reinforcement in Trachoma (HEAD START) is a surgical simulation device used to bridge the gap between classroom and live-surgery training specifically for trichiasis surgery. Long-term HEAD START practice will involve the following components, after completion of standard training (as described in the standard of care arm). Each week the participant will complete 2 surgeries on the HEAD START device. Monthly, the participant will send the accumulated cartridges to Addis Ababa for review by a senior trichiasis surgery trainer. The trainer will evaluate the cartridges and then will discuss his impression of the surgeries with the participant during a regular monthly call and note the findings. Practice will continue for 4-6 months, depending on the length of the rainy season and time of enrollment. At the end of the rainy season, an external examiner will evaluate the first 2 surgeries that the participant completes.
  Arms: Long-term HEAD START Training
Other: Standard of Care — All participants will receive trichiasis surgery training following Orbis' standard training approach, with the inclusion of HEAD START training between classroom and live surgery training. At the end of the surgical training session, an independent examiner will evaluate all trainees using the World Health Organization's Final Assessment of Surgeons form, as part of standard practice. The examiner also will complete a standard questionnaire focusing on the specific skill level achieved for each of the critical aspects of TT surgery. This form will be completed for all trainees undergoing training this spring, regardless of whether they are part of the long-term HEAD START assessment program.
  Arms: Standard of Care

SUMMARY:
The research group developed a surgical simulation device, the Human Eyelid Analogue Device for Surgical Training And skill Reinforcement in Trachoma (HEAD START), to bridge the gap between classroom and live-surgery training specifically for trichiasis surgery. In most settings, HEAD START is utilized once during training, then surgeons move on to live surgery and typically do not return to the simulator. The research team is interested in determining whether HEAD START provides benefit for long-term trichiasis surgery training, since many surgeons operate seasonally, with long periods of downtime between surgical camps and with little field supervision.

Participating surgeons will practice on HEAD START weekly, with monthly feedback from a senior supervisor. Researchers will assess their skill level at the start of HEAD START training and again at the start of the new surgical season in the fall of 2017. Researchers will also administer questionnaires to elicit feedback on the HEAD START training and supervision process.

DETAILED DESCRIPTION:
Eliminating blinding trachoma by 2020 is a key goal of the World Health Organization (WHO). Nearly 8 million individuals worldwide are in need of trichiasis surgery to prevent blindness.1 Currently, many trichiasis surgery programs experience poor outcomes in 10-50% of patients.2-11 High-quality surgery with minimal post-operative trichiasis is critical for success of the WHO goals. Typically, non-physician "surgeons" perform the procedure. Historically, they have been provided with one-week of classroom training and then begin live surgery training.

The research group developed a surgical simulation device, the Human Eyelid Analogue Device for Surgical Training And skill Reinforcement in Trachoma (HEAD START), to bridge the gap between classroom and live-surgery training specifically for trichiasis surgery. Based on this work, the WHO now recommends that all trainees receive training with a surgical simulation device before performing live surgery and that any refresher training should include simulation training as well.

In most settings, HEAD START is utilized once during training, meaning that once individuals are trained on HEAD START, they move on to live surgery and typically do not return to the simulator. In surgical sub-specialties with ready access to simulation devices, regular surgical simulation practice is utilized for skills maintenance and enhancement. The research team is interested in determining whether HEAD START provides benefit for long-term trichiasis surgery training, since many surgeons operate seasonally, with long periods of downtime between surgical camps and with little field supervision.

This project will compare skills of surgical trainees who continued with HEAD START practice and feedback throughout a 6-month break in surgery with those who did not. Study subjects will be selected based on their participation in an ORBIS-sponsored trichiasis surgery training program (either new training or refresher/conversion training). At the end of the standard training, the trainees who successfully complete training are ranked according to their scores on a classroom-based test and the WHO certification/assessment form. All individuals who successfully complete the training session and are scheduled to begin independent trichiasis surgery practice through the National Eye Care Program will be invited to participate in the study until we have reached 30 participants. Fifteen trainees will be invited to participate in long-term HEAD START practice in addition to performing regular live surgery. An additional 15 individuals will be selected for the trainer to assess their skill levels on live surgery at the end of training and again at the start of the surgical season this fall.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who have been selected to complete either

  1. new trichiasis surgery training through the Orbis Ethiopia of FHF training program OR
  2. refresher training for transitioning from bilamellar tarsal rotation surgery to posterior lamellar tarsal rotation surgery.
* Plans to continue practicing as a trichiasis surgeon throughout 2017.

Exclusion Criteria:

* Experienced surgeons who are retiring from surgical practice.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-05-17 (Actual); Primary Completion 2018-02-26 (Actual); Study Completion 2018-02-26 (Actual)

PRIMARY OUTCOMES:
Number of participants who feel long-term HEAD START use is beneficial for their surgical practice. | 6 months
  All participants and the senior trainers who conducted the monthly evaluations will be asked to complete an end of project questionnaire documenting their experience with HEAD START regarding the usefulness of regular surgical simulation practice, value of the monthly calls, and any recommendations for changes to the approach. Trainee and trainer responses to an end-of-project questionnaire regarding the utility of incorporating regular HEAD START practice will be analyzed to understand the benefit of regular HEAD START practice.

SECONDARY OUTCOMES:
Change in overall live-surgery training assessment scores between baseline and follow up | 6 months
  At the end of initial surgical trainings and again at the end of the rainy season, an independent examiner (not involved in the HEAD START evaluations) will assess the first 1-2 surgeries of the season of all study participants and all surgeons who successfully completed training in the spring but were not part of the long-term HEAD START assessment program. This assessment includes standard rankings of trainee skill.
Change in individual criterion scores for live surgery skills | 6 months
  At the end of initial surgical trainings and again at the end of the rainy season, an independent examiner (not involved in the HEAD START evaluations) will assess the first 1-2 surgeries of the season of all study participants and all surgeons who successfully completed training in the spring but were not part of the long-term HEAD START assessment program. This assessment includes standard rankings of trainee skill. Individual criterion scores for live surgery skills include incision placement and suturing placement, spacing and alignment
Change in individual criterion scores for live surgery skills among long-term HEAD START participants, comparing those who were the most highly active surgeons versus those who were the least active | 6 months
  Comparison in change in scores for individuals who were the most highly active surgeons versus those who were the least active but followed the HEAD START protocol.
  Surgeons will provide a record of the number of surgeries they completed each month (as part of standard practice). Criterion scores described in outcome 3 will be used to compare rates of change across level of surgical productivity (the number of surgeries performed).

CONTACTS AND LOCATIONS:
Overall Officials: Emily W Gower, Principal Investigator — University of North Carolina, Chapel Hill
Locations (3):
- Ethiopia (3):
  - Arbaminch Health Center, Gama Goffa, Southern Nations, Nationalities, and Peoples Region
  - Sodo Health Center, Wolaita, Southern Nations, Nationalities, and Peoples Region
  - Wolkite Health Center, Guragē, Southerns Nations, Nationalities, and Peoples Region

IPD SHARING:
Plan to Share IPD: No